CLINICAL TRIAL: NCT03984929
Title: Conexion: A Localized Information Resource on Diabetes and Depression for a Low-income Hispanic Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Rita Kukafka, Professor of Biomedical Informatics and Sociomedical Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAR5605; G08LM012689 (NIH)
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus; Depression
Keywords: Conexion; Diabetes; Depression; Low-income; Hispanic
MeSH Terms: conditions — Diabetes Mellitus; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Localized Information Resource Intervention (Experimental)
  Interventions: Behavioral: Conexion Localized
- Generic Information Resource Intervention (Active Comparator)
  Interventions: Behavioral: Conexion Generic

INTERVENTIONS:
Behavioral: Conexion Localized — The localized version of Conexion is an online health information resource on diabetes and depression tailored for the target community.
  Arms: Localized Information Resource Intervention
Behavioral: Conexion Generic — The generic version of Conexion is an online health information resource on diabetes and depression.
  Arms: Generic Information Resource Intervention

SUMMARY:
The proposed Conexion resource combines best publicly available evidence-based information and local community resources in one place. The information is curated and contextualized to meet local needs of consumers and providers. Content is tailored culturally and geographically to fit the community. This approach is consistent with evidence showing that individuals' interactions with health information and technology are "community embedded".

DETAILED DESCRIPTION:
Nationwide, Hispanics have many barriers to accessing health information, and are subject to significant health disparities, including disproportionate burden of diabetes and untreated mental illness. The research team's preliminary research has identified diabetes and depression as the highest priority needs in the study community of Washington Heights-Inwood (WAHI), which is an urban, low-income neighborhood in New York City with 71% Hispanic residents, predominantly immigrants from the Dominican Republic. Many high-quality health information resources already exist on the internet but they are not reaching many segments of the population, including parts of the WAHI community. The novel concept the investigators propose here is an information resource localized to a community.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Washington Heights/Inwood resident (zip codes 10032, 10033, 10034, 10040)
* interest in information on diabetes or depression
* speak English or Spanish

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Patient Activation | 1 month
  Person's active engagement in management of their own health will be measured as a patient activation measure (PAM) score. The PAM is a validated scale with 13 questions. The score ranges from 0 to 100, with a higher score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Kukafka, DrPH, FACMI, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Isabella Geriatric Center, New York, New York
  - YM-YWHA of Washington Heights, New York, New York